CLINICAL TRIAL: NCT06392685
Title: Clinical Performance of Repaired Resin Composite Restorations Using Separate Silane Coupling Agent Versus Adhesives Containing Regular or Acid Resistance Silane: A Randomized Controlled Trial
Brief Title: Composite Repair Using Silane Coupling Agent
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Fathy Talaat, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Composite repair
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Tooth Discoloration; Hypersensitivity; Tooth Fracture; Dental Restoration Failure of Marginal Integrity
Keywords: Silane coupling agent; Adhesive containing silane; Acid resistance silane containing adhesive.; Defective resin composite restoration; Repair of posterior resin composite
MeSH Terms: conditions — Tooth Discoloration; Hypersensitivity; Tooth Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Silane coupling agent(Comparator) (Active Comparator): In the control group, Silane coupling agent (Porcelain primer) will be applied following the acid etch rinsing and drying step, for 30 seconds and then it will be thoroughly dried using air syringe then universal adhesive with regular silane will be actively applied for 20 seconds and then it will be light cured for 20 seconds and final restoration will be done.
  Interventions: Other: Silane coupling agent
- .Adhesive containing silane.(Intervention 1 ) (Active Comparator): Universal adhesive with regular silane will be applied for 20 seconds, air thinned for 10 seconds and then it will be light cured for 20 seconds and final restoration will be done using same resin composite material
  Interventions: Other: Adhesive containing silane.(Intervention 1 )
- Acid resistance silane containing adhesive.(Intervention 2) (Active Comparator): Acid resistance silane containing adhesive will be applied for 20 seconds, dry with gentle air for 3 seconds, then with stronger air and light cured for 10 seconds and final restoration will be done
  Interventions: Other: Acid resistance silane containing adhesive.(Intervention 2)

INTERVENTIONS:
Other: Silane coupling agent — Silane coupling agent (Porcelain primer) will be applied following the acid etch rinsing and drying step, for 30 seconds and then it will be thoroughly dried using air syringe then universal adhesive with regular silane will be actively applied for 20 seconds and then it will be light cured for 20 seconds and final restoration will be done
  Arms: Silane coupling agent(Comparator)
Other: Adhesive containing silane.(Intervention 1 ) — Universal adhesive with regular silane will be applied for 20 seconds, air thinned for 10 seconds and then it will be light cured for 20 seconds and final restoration will be done using same resin composite material
  Arms: .Adhesive containing silane.(Intervention 1 )
Other: Acid resistance silane containing adhesive.(Intervention 2) — Acid resistance silane containing adhesive will be applied for 20 seconds, dry with gentle air for 3 seconds, then with stronger air and light cured for 10 seconds and final restoration will be done
  Arms: Acid resistance silane containing adhesive.(Intervention 2)

SUMMARY:
Evaluation the influence of the use of silane coupling agent application as a separate step versus application of silane or acid resistance silane containing adhesives on the clinical performance of repaired posterior resin composite restorations according to Modified United States Public Health Service (USPHS) criteria over one year.

DETAILED DESCRIPTION:
some manufacturers have produced silane-containing adhesives in their new products, which might eliminate the need to apply separate silane. However, this silane coupling agent can be hydrolyzed by the acidic monomer in the adhesive making it useless. Acid resistance silane containing adhesive is the update version of the silane containing adhesive which provides a long lasting effective bond between the old and new resin composite restorations

ELIGIBILITY:
Inclusion Criteria:

* Participants Inclusion:

Patients aging (18-45). Patients with a high level of oral hygiene. Patients with good likelihood of recall availability. - Teeth Inclusion: The restorations were first placed 12 to 24 months ago. Teeth with healthy remaining tooth structure. Posterior restorations with approximately 3mm in size occlusal marginal defect. Asymptomatic teeth before repair.

Exclusion Criteria:

* Participants Exclusion:

Patient with high caries risk Patient with poor periodontal health. Heavy bruxism habits. Pregnant or lactating females.

-Teeth Exclusion: The restorations with large defects The restorations in the third molars Last experience with allergic reactions against any components of the used materials.

Patients receiving orthodontic treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation | T0= Baseline 24 hours postoperative. T1= 6 months follow up. T2= 12 months follow up.
  Alpha (A) Restoration adapts closely to the tooth structure; there is no visible crevice Bravo (B) There is a visible crevice, the explorer will penetrate, without dentin exposure.
  Charlie(C) The explorer penetrates into a crevice in which dentin or the base is exposed.

SECONDARY OUTCOMES:
Anatomical form | T0= Baseline 24 hours postoperative. T1= 6 months follow up. T2= 12 months follow up.
  Alpha (A)Anatomic form ideal Bravo (B)Restoration is under contoured, without dentin, or base exposure Charlie (C)Restoration is under contoured, with dentin or base exposure; anatomic form is unsatisfactory; restoration needs replacement
Marginal discoloration | T0= Baseline 24 hours postoperative. T1= 6 months follow up. T2= 12 months follow up.
  Alpha(A) No marginal discoloration. Bravo(B)Minor marginal discoloration without staining toward the pulp, only visible using a mirror and operating light. Charlie(C) Deep discoloration with staining toward the pulp, visible at a speaking distance of 60 to 100 cm.
Surface roughness | T0= Baseline 24 hours postoperative. T1= 6 months follow up. T2= 12 months follow up.
  Alpha(A) As smooth as the surrounding enamel. Bravo(B) Rougher than surrounding enamel; improvement by finishing is feasible Charlie(C) Very rough, could become anti-esthetic and/or retain biofilm; improvement by finishing is not feasible
Secondary caries | T0= Baseline 24 hours postoperative. T1= 6 months follow up. T2= 12 months follow up.
  Alpha :No active caries present Charlie: Active caries is present in contact with the restoration
Postoperative sensitivity | T0= Baseline 24 hours postoperative. T1= 6 months follow up. T2= 12 months follow up
  Alpha :No postoperative sensitivity Charlie: Short-term and tolerable postoperative sensitivity